CLINICAL TRIAL: NCT03940339
Title: Effect of Suboccipital Muscle Myofascial Release on Hamstring Muscle Length, Pain and Disability in Patients With Anterolisthesis
Brief Title: Suboccipitalis Myofascial Release in Hamstring Tightness in Patients With Anterolisthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 lockdown
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Supervisor and Associate Professor, Department of Pediatric and Neonatal Physiotherapy, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDU/IEC/1369; U1111-1232-1359 (Other: UTN by WHO International Clinical Trial Registry Platform)
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Anterolisthesis
Keywords: Hamstring muscles; Pain measurement; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Two group pretest posttest randomized control design
Who Masked: Participant
Masking Description: Single blinded participants will be recruited
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital myofascial release (Experimental): Treatment will be given for 3 minutes, 3 days per week for 4 weeks.
  Interventions: Other: Suboccipital myofascial release
- Coventional Physiotherapy (Active Comparator): Treatment will be given for 3 days per week for 4 weeks
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Suboccipital myofascial release — The MFR technique will be given in the upper cervical region with the patient in supine position. The MFR will be given for three repetitions per session, three times per week for the period of four weeks.
  Arms: Suboccipital myofascial release
Other: Conventional Physiotherapy — The control group will be receiving conventional physiotherapy treatment for hamstring tightness which includes static stretching, modified hold-relax stretching and contract relax technique.
  Arms: Coventional Physiotherapy

SUMMARY:
Background:

Anterolisthesis presents with tightness of hamstring muscle which is a major contributing factor for low back pain and disability. Suboccipital Myofascial release decreases the tension in the fascia and helps to amend the muscle imbalance. There is a presence of superficial backline between suboccipitalis and hamstring muscle.

Aim:

The purpose of the study is to find out the effect of sub occipital myofascial release on hamstring tightness along with pain and disability associated with it in Anterolisthesis.

Methods:

The study will recruit individuals with Anterolisthesis between the age of 35- 55. Pathologies which will limit or interfere with the test outcome shall be excluded. The samples will be collected using criterion based sampling. Procedure will be explained prior to the intervention

Data analysis:

Normality of the collected data will be established by Shapiro Wilk Test. Based on the normality, descriptive statistics data will be expressed as mean ± standard deviation or median and intra quartile range. Within group comparison will be done by paired t test or Wilcoxon signed rank test and between group comparison will be done through independent t test or Mann Whitney U test.

DETAILED DESCRIPTION:
1. Introduction:

   Anterolisthesis refers to an anterior displacement of a vertebra over subjacent vertebra causing low back pain, radiculopathy and hamstring tightness. Hamstring tightness causes improper patterns in the lumbopelvic region. There is a dura matter which connects suboccipitalis and hamstring muscle and reduction in the tone of suboccipitalis will thus cause decrease in tone of hamstring muscle. Myofascial release is a manipulative treatment that attempts to release tension in fascia and has an effect to decrease soreness of muscle.

   1.1.Problem statement: Generally in patients with anterolisthesis a single component is considered as a treatment, this study thus aims to be a bridge filling the gap in the scientific cognizance

   1.2.Purpose of the study:The target of the study is to see the outcome of sub occipitalis myofascial release on tightness of hamstring muscle, pain and disability.

   1.3.Objectives of the study: To evaluate the efficacy of suboccipital myofascial release and conventional physiotherapy treatment in tightness of hamstring muscle, pain and disability
2. Procedure:

Total male (n) and female (n) patients between the age of 35 and 55 years with grade 1 and 2 Anterolisthesis will be selected on the basis of inclusion and exclusion criteria. The suitable sample will be randomly allocated into 2 groups - experimental and control group respectively. The popliteal angle test will be carried out to assess hamstring length and modified oswestry disability index will be used to quantify disability for low back pain. Visual analogue scale will be used to measure intensity of pain. All the necessary measures will be taken among the participants of experimental group.The MFR technique will be given in the upper cervical region with the patient in supine position. The MFR will be given for three repetitions per session, three times per week for the period of four weeks. The control group will be receiving conventional physiotherapy treatment for hamstring tightness which includes static stretching, modified hold-relax stretching and contract relax technique.

ELIGIBILITY:
Inclusion criteria:

Patients aged between 35-55 years Both male and female Individuals with Hamstring tightness Individual with Anterolisthesis Individual with pain and disability

Exclusion Criteria:

Individuals with neck pain Patients with history of neck trauma Fracture of lower limb Cervical ligament instability Spinal fractures in the past 6 months Open wounds and skin allergies in the back

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Popliteal Angle Test | 2 weeks
  Popliteal angle is an assessment of the tone of the hamstring muscles. The thigh is flexed on the abdomen with one hand and then the other hand straightens the leg by pushing on the back of the ankle until there is firm resistance to the movement. Popliteal angle is measured in degrees.
Modified Oswerstry Disability Index | 2 weeks
  It is an extremely important tool used to measure a patient's permanent functional disability. The total score range from 0-50.

SECONDARY OUTCOMES:
Visual Analogue Scale | 2 weeks
  It is a quantifying instrument for subjective characteristics or attitudes of pain that cannot be directly measured. The total score range from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Bishaka Pradhan, BPT, (MPT), Principal Investigator — Department of Musculoskeletal Physiotherapy, MMIPR
Locations (1):
- Maharishi Markandeshwar Hospital, Mullana, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No
It is not yet decided

REFERENCES:
- [Result] Vatsal DK, Kainth R, Kainth R, Husain PM. Original Article A clinico-etiological study of spondylolisthesis in north Indian population. Int J Med Sci Clin Invent. 2017;4(5):2884-7.